CLINICAL TRIAL: NCT05168384
Title: Randomized, Controlled, Open-label Study Evaluating the Safety and Efficacy of Extracorporeal Photopheresis (ECP) in the Treatment of Multiple Sclerosis
Brief Title: Safety and Efficacy of Extracorporeal Photopheresis (ECP) in the Treatment of Multiple Sclerosis
Acronym: PHOMS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abu Dhabi Stem Cells Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT.005.2.0.PHOMS; DOH/CVDC/2022/155 (Other: Abu Dhabi Health Research and Technology Ethics Committee (ADHRTC))
Record Dates: First submitted 2021-11-25; First posted 2021-12-23 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive
Keywords: Extracorporeal Photopheresis; Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Photopheresis; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (ECP + SoC Group) (Experimental): Extracorporeal photopheresis (ECP) plus Multiple Sclerosis (MS) standard of care
  Interventions: Combination Product: Extracorporeal Photopheresis; Combination Product: MS standard of care
- Group B (SoC Group) (Active Comparator): MS standard of care alone (SoC, defined by Disease-modifying Therapy -DMT, recommended by the American Academy of Neurology -AAN
  Interventions: Combination Product: MS standard of care

INTERVENTIONS:
Combination Product: Extracorporeal Photopheresis — ECP procedures will be performed using a Therakos Cellex integrated, closed photopheresis system (Therakos, Inc., a Mallinckrodt Pharmaceuticals Company).
  ECP will administered according to the following schedule (Group A):
  Weeks 1-8: Twice per week (16 sessions). Weeks 9-16: Once per week (8 sessions). Weeks 17-24: Once every 2 weeks (4 sessions). Total: 28 sessions (within 24 weeks).
  Other Names: Extracorporeal Photoimmunotherapy; Photochemotherapy
  Arms: Group A (ECP + SoC Group)
Combination Product: MS standard of care — Disease-modifying Therapy -DMT, recommended by the American Academy of Neurology -AAN
  Other Names: Disease-modifying Therapies

SUMMARY:
PHOMS Study is a randomized, controlled, open-label, prospective, and multicentric clinical trial involving outpatients diagnosed with Secondary Progressive Multiple Sclerosis (SPMS) or Relapsing-Remitting Multiple Sclerosis (RRMS). The primary objective is the safety profile assessment of the investigational intervention (Extracorporeal Photopheresis -ECP) and its preliminary efficacy evaluation, while the secondary objective is the assessment of the immune response profile in MS patients.

DETAILED DESCRIPTION:
PHOMS patients will be randomly allocated (2:1) in a parallel assignment involving two groups of participants: Group A (Experimental group, n = 30): ECP plus Multiple Sclerosis (MS) standard of care, or Group B (Control group, n = 15) receiving MS standard of care alone. The PHOMS Study standard of care is defined by Disease-modifying Therapy (DMT) recommended by the American Academy of Neurology (AAN). The Study will be conducted within Abu Dhabi Stem Cells Center (ADSCC) and Yas Clinic Khalifa City (YCKC) Hospital, including patient assessment and inclusion, randomization, ECP procedures (Group A), and follow-up consultations, according to the approved Protocol and Good Clinical Practices (GCPs) principles. The primary objective is the safety profile assessment of the investigational intervention (ECP), to be assessed by procedure tolerability, the incidence of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0), and the World Health Organization - Uppsala Monitoring Center (WHO-UMC) causality assessment system. The ECP preliminary efficacy assessment, as another primary objective, will be assessed by the proportion of subjects with no evidence of disease progression at 1 year; while the secondary objective is the assessment of the immune response profile in MS patients. All subjects will undergo longitudinal Expanded Disability Status Scale (EDSS), 25-foot walk ambulation test, 9-hole peg test, and 36-Item Short Form Survey (SF-36) testing at baseline and every 3 months through 1 year. Blood will be collected for immunological testing at baseline, months 3, 6, 9, and 12; and subjects will also undergo neuroimaging with brain Magnetic Resonance Imaging (MRI) at baseline, and months 6 and 12 following initiation of treatment, while Chest X-Ray, electrocardiogram (ECG), and echocardiogram can be required at the discretion of the Investigator. The trial is approved by the institutional Research Ethics Committees (RECs), and written informed consent will be obtained from all patients. PHOMS Study will be conducted following the principles of the Declaration of Helsinki and the International Conference on Harmonization (ICH) GCP Guidelines. The authors are responsible for designing the trial and for compiling and analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrate Expanded Disability Status Scale (EDSS) scores between 3 to 6.5 at screening.
2. Documented EDSS progression in the 2 years prior to screening of 1 point or greater for patients with an EDSS score less than 6 at baseline, and greater than or equal to 0.5 for patients with an EDSS score greater than or equal to 6.0 at baseline *.

   * If documented EDSS scores are not available, a written summary of the clinical evidence of disability progression over the last 2 years, and retrospective assessment of EDSS score from data in the medical records, must be submitted for review by the principal investigators.
3. Documented initial onset characterized by a relapsing-remitting course as described in the Diagnostic Criteria.
4. Age ≥ 18 ≤ 75 years.
5. Weight > 40 kg.
6. Hematocrit ≥ 28 % (with or without transfusion support).
7. Platelet count > 100,000 per μL (with or without transfusion support).
8. Willingness to use at least 1 reliable method of birth control (e.g., abstinence, oral contraceptives, intrauterine devices, barrier method with spermicide, or surgical sterilization) throughout the study for all men and women of childbearing potential.
9. Willingness to participate in all PHOMS Study tests, visits, and procedures (including the ECP), as outlined in the informed consent.
10. Patients must have adequate peripheral venous access to initiate ECP therapy, and central line insertion shall be required.
11. The patient agrees to participate in the trial and signs the PHOMS Study informed consent form.

Exclusion Criteria:

1. Absolute medical contraindication to receive ECP.
2. Laboratory evidence of any of the following:

   * White blood cells (WBC) < 2,000 cells per uL.
   * Serum transaminase levels > x 2 UNL.
   * Creatinine Clearance < 60 mL/min.
3. Concurrent diagnosis of a neurological condition that would interfere with the assessment of MS, or an autoimmune disease or inflammatory condition that is chronically treated with immunosuppressive agents.
4. Evidence of known infection with human immunodeficiency virus (HIV) or active (not including latent) Hepatitis B.
5. Uncontrolled infection requiring treatment at study entry.
6. Hypersensitivity or allergy to psoralen (methoxalen).
7. Hypersensitivity or allergy to both heparin and citrate products (If hypersensitive or allergic to only one of these products, exclusion does not apply).
8. Inability to tolerate fluid changes associated with ECP (e.g., inadequate renal, hepatic, pulmonary and cardiac function leading to enable patient to tolerate extracorporeal volume shifts associated with ECP).
9. Presence of aphakia or photosensitive disease (systemic lupus erythematosus, porphyrias, etc.).
10. Women who are pregnant and/or lactating.
11. Use of any investigational drug/treatment at the time of enrollment or within the previous 60 days, or five elimination half-lives, or until the expected pharmodynamic effect has returned to baseline, whichever is longer.
12. Treatment with any of the medications or procedures listed below:

    * Natalizumab, or rituximab within 3 months prior to randomization.
    * Cyclophosphamide within 1 year prior to randomization.
    * Mitoxantrone, ofatumumab, ocrelizumab, cladribine, or daclizumab within 1 years prior to randomization.
    * Intravenous immunoglobulin within 3 months prior to randomization.
    * Plasmapheresis within 3 months prior to randomization.
13. Inability to undergo MRI scans.
14. Contraindication to gadolinium due to past allergic, hypersensitive, or adverse reaction or impaired renal function. Patients receiving a steroid prep prior to gadolinium administration due to history of hypersensitivity or allergy to other agents or due to prior mild reaction to gadolinium will not be excluded from the study.
15. Poor venous access.
16. Previous history of skin cancer, leukemia / lymphoma / myeloma, or bone marrow transplant.
17. Patients taking Coumadin who are unable to switch from oral anticoagulants to enoxaparin.
18. Heparin-induced thrombocytopenia.
19. Poor cardiac function.
20. Severe hypotension.
21. Any other disease or condition which, in the opinion of the investigator, could interfere with participation according to the PHOMS Study Protocol, or with the ability of the patients to cooperate and comply with study procedures.
22. Inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-26 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tolerability to ECP procedures (Group A patients) | Weeks 0-24
  Proportion of patients tolerating the ECP procedures reaching the cycles' goal.
Incidence of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) | Weeks 0-52
  Proportion of patients referring TEAEs, AESIs, and SAEs assessed by CTCAE v5.0.
Tolerability to TEAEs, AESIs, and SAEs | Weeks 0-52
  Proportion of patients tolerating TEAEs, AESIs, and SAEs, and finalizing the Study
Clinical improvement (25-foot walk) | Baseline, months 3, 6, 9, and 12
  Proportion of patients with clinical improvement from baseline in 20% or greater increase in the timed 25-foot walk
Clinical improvement (9-hole peg test) | Baseline, months 3, 6, 9, and 12
  Proportion of patients with clinical improvement from baseline in 20% or greater increase in the 9-hole peg test
Clinical improvement (36-Item Short Form Survey) | Baseline, months 3, 6, 9, and 12
  Proportion of patients with clinical improvement from baseline in 20% or greater increase in the 36-Item Short Form Survey (SF-36)
Clinical improvement (EDSS baseline low score) | Baseline, months 3, 6, 9, and 12
  Proportion of patients with clinical improvement from baseline in 1 point or greater increase in EDSS score (in subjects with baseline EDSS scores between 3 and 5.5)
Clinical improvement (EDSS baseline high score) | Baseline, months 3, 6, 9, and 12
  Proportion of patients with clinical improvement from baseline in 0.5 point or greater increase in EDSS score (in subjects with baseline EDSS scores ≥ than 6)
Occurrence of clinical relapse at any point in the study | Weeks 0-52
  Proportion of patients demonstrating new or recurrent neurological symptoms consistent with MS, symptoms last 24 to 48 hours, or development of new MS symptoms over days to weeks

SECONDARY OUTCOMES:
Immune response profile (cellular) | Baseline, months 3, 6, 9, and 12
  Analysis of the biomarkers CD3, CD4, CD8, CD11c, CD14, CD16, CD19, CD20, CD25, CD27, CD28, CD38, CD45, CD45RA, CD45RO, CD56, CD57, CD66b, CD123, CD127, CD161, CD294, CCR4, CCR6, CCR7, CXCR3, CXCR5, for identification of immune cells and subsets analysis
Immune response profile (humoral) | Baseline, months 3, 6, 9, and 12
  IgG, IgA, IgM levels will be assessed for characterization of the humoral response profile

CONTACTS AND LOCATIONS:
Overall Officials: Yendry Ventura Carmenate, M.D., Principal Investigator — Abu Dhabi Stem Cells Center
Locations (1):
- Abu Dhabi Stem Cells Center, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castillo-Aleman YM, Villegas-Valverde CA, Ventura-Carmenate Y, Al-Kaabi FM, Lumame S, Castelo C, Mir R, Brylev L, Atieh M, Haider MT, Bencomo-Hernandez AA. Mononuclear cell recruitment during extracorporeal photopheresis: Partial results of a phase 1/2 randomized clinical trial in multiple sclerosis. Transfus Apher Sci. 2025 Apr;64(2):104095. doi: 10.1016/j.transci.2025.104095. Epub 2025 Feb 9. PMID 39947046
- [Background] Castillo-Aleman YM, Lumame S, Castelo C, Mir R, Ventura-Carmenate Y, Al-Kaabi FM. Recurrent clumping in the extracorporeal photopheresis circuit using acid citrate dextrose solution A. J Clin Apher. 2024 Jun;39(3):e22117. doi: 10.1002/jca.22117. No abstract available. PMID 38661254